CLINICAL TRIAL: NCT03915132
Title: Phase II Trial of Nimotuzumab Combined With Volumetric Modulated Arc Therapy in Elderly Patients With Nasopharyngeal Carcinoma
Brief Title: Nimotuzumab Combined With VMAT in Elderly Patients With Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun-Lin Yi, MD, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1937
Record Dates: First submitted 2019-03-31; First posted 2019-04-16 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: VMAT; Nimotuzumab; Elderly Patients; efficacy; toxicity
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VMAT plus Nimotuzumab (Experimental): Patients receive Nimotuzumab weekly during radiotherapy .
  Interventions: Drug: Nimotuzumab; Radiation: VMAT

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 200mg/m2 IV on d1 of a week before radiotherapy , and 100mg/m2 IV on d1 weekly for 7 cycles
  Other Names: Taixinsheng
Radiation: VMAT — Intensity-modulated radiotherapy was given to the patients with regimen of 69.96 Gy-73.92 Gy to the gross target volume of nasopharynx,69.96 Gy to the gross target volume of positive nodes, 60.06 Gy the high risk clinical target volume, 50.96 Gy to the low risk clinical target volume.

SUMMARY:
To evaluate the efficacy and toxicity of Nimotuzumab combined with VMAT in the treatment of elderly patients with nasopharyngeal carcinoma (> 70 years old), and to provide high-level clinical evidence for the optimal treatment of elderly patients with nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
The incidence of elderly patients with nasopharyngeal carcinoma is increasing with a rapidly ageing population. However, the prognosis is worse than that of young patients. Some patients can benefit from intensive treatment such as concurrent chemoradiotherapy, but are always with obvious toxicity. With the advancement of radiotherapy technology and the emergence of molecular targeted drugs, radiotherapy combined with Nimotuzumab has shown good therapeutic efficacy and tolerance. The investigators plan to testify VMAT combined with Nimotuzumab in elderly patients with nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed squamous cell carcinoma of nasopharynx; Aged ≥ 70 years old; Stage III-IVB diseases according to 8th AJCC Staging; Treatment for the first time; ECOG scores ≤ 1; Normal hepatic, renal and bone-marrow function; ACE-27 scores ≤2; Life expectancy≥12 weeks; Can understand and sign the consent.

Exclusion Criteria:

* Past malignancies history (except for non-melanoma skin cancer or cervical carcinoma in situ or cured prostate cancer of early stage); Allergic to Nimotuzumab; Severe comorbidities including cardiovascular, cerebral vascular, mental and uncontrolled diabetes disease; Chemotherapy, surgery or other molecule-target treatment; Severe malnutrition.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 4 months
  Complete remission rate will be measured by RECIST 1.1

SECONDARY OUTCOMES:
acute treatment toxicity | up to 16 weeks
  Acute toxicity will be measured by CTCAE4.0
Quality of Life Assessment | 2 years
  EORTC,QLQ-C30 Version 3.0 are used.
local control rate | 2 years
regional control rate | 2 years
late treatment toxicity | 2 years
  late toxicity will be measured by CTCAE4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, professor, Principal Investigator — CAMS
Locations (1):
- Cancer hospital, Chinese Academy of Medical Sciences, Beijin, China

REFERENCES:
- [Background] Cao C, Hu Q, Chen X. Intensity-modulated radiotherapy for elderly patients with nasopharyngeal carcinoma. Head Neck. 2018 Mar;40(3):590-595. doi: 10.1002/hed.25016. Epub 2017 Nov 20. PMID 29155480
- [Background] Liu H, Chen QY, Guo L, Tang LQ, Mo HY, Zhong ZL, Huang PY, Luo DH, Sun R, Guo X, Cao KJ, Hong MH, Mai HQ. Feasibility and efficacy of chemoradiotherapy for elderly patients with locoregionally advanced nasopharyngeal carcinoma: results from a matched cohort analysis. Radiat Oncol. 2013 Mar 22;8:70. doi: 10.1186/1748-717X-8-70. PMID 23521779
- [Result] Zhang Y, Yi JL, Huang XD, Xu GZ, Xiao JP, Li SY, Luo JW, Zhang SP, Wang K, Qu Y, Gao L. Inherently poor survival of elderly patients with nasopharyngeal carcinoma. Head Neck. 2015 Jun;37(6):771-6. doi: 10.1002/hed.23497. Epub 2015 Feb 11. PMID 24115004
- [Result] Jin YN, Zhang WJ, Cai XY, Li MS, Lawrence WR, Wang SY, Mai DM, Du YY, Luo DH, Mo HY. The Characteristics and Survival Outcomes in Patients Aged 70 Years and Older with Nasopharyngeal Carcinoma in the Intensity-Modulated Radiotherapy Era. Cancer Res Treat. 2019 Jan;51(1):34-42. doi: 10.4143/crt.2017.551. Epub 2018 Feb 6. PMID 29409313